CLINICAL TRIAL: NCT01393613
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Fixed-dose OPC-34712 in the Treatment of Adults With Acute Schizophrenia
Brief Title: Efficacy Study of OPC-34712 in Adults With Acute Schizophrenia
Acronym: BEACON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-10-230
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Acute Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 3 OPC 34712 (Experimental): Higher dose, tablet, once daily, for six weeks
  Interventions: Drug: OPC-34712
- Dose 2 OPC 34712 (Experimental): Middle dose, tablet, once daily, for six weeks
  Interventions: Drug: OPC-34712
- Dose 1 OPC 34712 (Experimental): Lower dose, tablet, once daily, for six weeks
  Interventions: Drug: OPC-34712
- Placebo (Placebo Comparator): Placebo, once daily, for six weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-34712 — Higher dose tablet, once daily, for six weeks,
  Arms: Dose 3 OPC 34712
Drug: OPC-34712 — Middle dose tablet, once daily, for six weeks
  Arms: Dose 2 OPC 34712
Drug: OPC-34712 — Lower dose tablet, once daily, for six weeks
  Arms: Dose 1 OPC 34712
Drug: Placebo — Placebo, once daily, for six weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of fixed doses of OPC-34712 versus placebo for the treatment of adult subjects with an acute relapse of schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely debilitating mental illness that affects approximately 1% of the world population. Hallucinations and delusions are the most striking characteristic positive symptoms of schizophrenia; however, more subtle negative symptoms (eg, social withdrawal and lack of emotion, energy, and motivation) may also be present. The first antipsychotics developed for the treatment of schizophrenia were effective against positive symptoms, but showed little efficacy for negative symptoms and were also associated with a high incidence of side effects. Second generation antipsychotics, represent a significant advancement in the treatment of psychotic disorders because they are effective and at the same time exhibit fewer side effects than first generation antipsychotics. Although generally safer than first generation antipsychotics, the second-generation antipsychotics are not devoid of undesirable side effects such as Hyperprolactinemia and weight gain. In addition, the safety of these drugs vary considerably.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years of age, with a diagnosis of schizophrenia, as defined by DSM-IV-TR criteria
2. Subjects who have been recently hospitalized or who would benefit from hospitalization for an acute relapse of schizophrenia
3. Subjects experiencing an acute exacerbation of psychotic symptoms
4. Other protocol specific inclusion criteria may apply

Exclusion Criteria:

1. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug
2. Subjects with a current DSM-IV-TR Axis I diagnosis of:

   * Schizoaffective disorder
   * MDD
   * Bipolar disorder
   * Delirium, dementia, amnestic or other cognitive disorder
   * Borderline, paranoid, histrionic, schizotypal, schizoid or antisocial personality disorder
3. Subjects presenting with a first episode of schizophrenia
4. Other protocol specific exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Skuban, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (53):
- United States (18):
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - Escondido, California
  - Long Beach, California
  - Orange, California
  - Pico Rivera, California
  - San Diego, California
  - North Miami, Florida
  - Overland Park, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - St Louis, Missouri
  - Buffalo, New York
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
- Colombia (3):
  - Bogotá
  - Medellín
  - Pereira
- Croatia (2):
  - Rijeka
  - Zagreb
- Mexico (5):
  - Col. Florida, Mexico City
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potos
  - Monterrey
- Philippines (5):
  - Cebu City
  - Davano City
  - Makati City
  - Mandaluyong
  - Manila
- Russia (10):
  - Arkhangelsk
  - Moscow
  - Moscow Region
  - Nizhny Novgorod
  - Petrozavodsk
  - Saint Petersburg
  - Samara
  - Saratov
  - Tomsk
  - Village Nikolskoe
- Slovakia (5):
  - Bojnice
  - Bratislava
  - Michalovace
  - Rimavská Sobota
  - Rožňava
- Taiwan (5):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Ismail Z, Kapadia S, Palma AM, Yildirim M, Farovik A. Brexpiprazole for anxiety symptoms in schizophrenia: a pooled analysis of short- and long-term trials. Curr Med Res Opin. 2025 Aug;41(8):1535-1548. doi: 10.1080/03007995.2025.2552286. Epub 2025 Sep 11. PMID 40859756
- [Derived] Ismail Z, Meehan SR, Farovik A, Kapadia S, Palma AM, Zhang Z, McIntyre RS. Effects of brexpiprazole on patient life engagement in schizophrenia: post hoc analysis of Positive and Negative Syndrome Scale data. Curr Med Res Opin. 2025 Jan;41(1):145-153. doi: 10.1080/03007995.2024.2440059. Epub 2025 Jan 3. PMID 39749727
- [Derived] Correll CU, He Y, Therrien F, MacKenzie E, Meehan SR, Weiss C, Hefting N, Hobart M. Effects of Brexpiprazole on Functioning in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. J Clin Psychiatry. 2022 Mar 1;83(2):20m13793. doi: 10.4088/JCP.20m13793. PMID 35235720
- [Derived] Marder SR, Meehan SR, Weiss C, Chen D, Hobart M, Hefting N. Effects of Brexpiprazole Across Symptom Domains in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. Schizophr Bull Open. 2021 May 1;2(1):sgab014. doi: 10.1093/schizbullopen/sgab014. eCollection 2021 Jan. PMID 34901863
- [Derived] Newcomer JW, Eriksson H, Zhang P, Weiller E, Weiss C. Changes in metabolic parameters and body weight in brexpiprazole-treated patients with acute schizophrenia: pooled analyses of phase 3 clinical studies. Curr Med Res Opin. 2018 Dec;34(12):2197-2205. doi: 10.1080/03007995.2018.1498779. Epub 2018 Jul 27. PMID 29985680
- [Derived] Kane JM, Skuban A, Hobart M, Ouyang J, Weiller E, Weiss C, Correll CU. Overview of short- and long-term tolerability and safety of brexpiprazole in patients with schizophrenia. Schizophr Res. 2016 Jul;174(1-3):93-98. doi: 10.1016/j.schres.2016.04.013. Epub 2016 May 14. PMID 27188270
- [Derived] Kane JM, Skuban A, Ouyang J, Hobart M, Pfister S, McQuade RD, Nyilas M, Carson WH, Sanchez R, Eriksson H. A multicenter, randomized, double-blind, controlled phase 3 trial of fixed-dose brexpiprazole for the treatment of adults with acute schizophrenia. Schizophr Res. 2015 May;164(1-3):127-35. doi: 10.1016/j.schres.2015.01.038. Epub 2015 Feb 12. PMID 25682550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 674 participants from 68 trial sites in 8 countries.
Pre-assignment Details: Adults with schizophrenia as defined by Diagnostic and Statistical Manual of Mental Health Disorders 4th Edition Text Revision criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) for schizophrenia and psychotic disorders studies were included.
Groups:
- Brexpiprazole 1 mg: Brexpiprazole 1 mg tablet once daily for 6 weeks.
- Brexpiprazole 2 mg: Brexpiprazole 2 mg tablet once daily for 6 weeks.
- Brexpiprazole 4 mg: Brexpiprazole 4 mg tablet once daily for 6 weeks.
- Placebo: Placebo tablet once daily for 6 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Started | 120 | 186 | 184 | 184
Completed | 81 | 129 | 130 | 118
Not Completed | 39 | 57 | 54 | 66
Not completed — Adverse Event | 11 | 11 | 13 | 22
Not completed — Participant Met Withdrawal Criteria | 0 | 0 | 2 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 15 | 25 | 23 | 21
Not completed — Protocol Deviation | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 9 | 20 | 16 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo | Total
Number analyzed (Participants) | 120 | 186 | 184 | 184 | 674
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (11.9) | 36.9 (10.9) | 38.6 (11.0) | 39.3 (10.8) | 38.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 64 | 71 | 73 | 251
  Male | 77 | 122 | 113 | 111 | 423

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: Efficacy sample consisted of all participants who received at least one dose of study medication and have Baseline and at least one Post-Baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -3.32 (0.83) | -4.35 (0.68) | -5.58 (0.68) | -3.48 (0.68)
  Week 2 | -7.61 (1.09) | -8.70 (0.88) | -8.42 (0.88) | -6.61 (0.89)
  Week 3 | -11.56 (1.30) | -10.69 (1.06) | -12.63 (1.05) | -8.95 (1.06)
  Week 4 | -13.97 (1.49) | -13.12 (1.21) | -15.55 (1.19) | -11.10 (1.22)
  Week 5 | -14.47 (1.71) | -14.11 (1.38) | -17.26 (1.37) | -11.89 (1.40)
  Week 6 | -16.90 (1.86) | -16.61 (1.49) | -20.00 (1.48) | -13.53 (1.52)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare the average effect analysis for brexpiprazole 2 mg/day and 4 mg/day and placebo combined treatment groups at Week 6. The primary analysis was performed by fitting a Mixed Model Repeated Measures (MMRM) with an unstructured variance covariance structure. The model included fixed class effect terms for treatment, trial site, visit week, baseline, baseline and visit interaction and an interaction term of treatment by visit week; Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; MMRM analysis fixed effect of treatment, trial site, visit, treatment visit interaction, Baseline value, Baseline visit interaction as covariates
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.47, 95% CI 2-sided [-10.6 to -2.35]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1448, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.08, 95% CI 2-sided [-7.23 to 1.07]
Statistical Analysis 4: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6. MMRM analysis fixed effect of treatment, clinical visit, trial site, treatment visit interaction, Baseline value, and Baseline visit interaction as covariates; Test type: Superiority or Other; p = 0.1588, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.37, 95% CI 2-sided [-8.06 to 1.32]

2. Secondary Outcome: Mean Change From Baseline to Week 6 in Clinical Global Impression-Severity (CGI-S) Score.
Description: Severity of illness for each participant was rated using the CGI-S, which was the key secondary efficacy endpoint. To perform this assessment, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 120 | 180 | 183 | 181
Units on a scale
  Week 1 | -0.11 (0.05) | -0.16 (0.04) | -0.22 (0.04) | -0.12 (0.04)
  Week 2 | -0.31 (0.06) | -0.40 (0.05) | -0.40 (0.05) | -0.36 (0.05)
  Week 3 | -0.63 (0.07) | -0.60 (0.06) | -0.69 (0.06) | -0.44 (0.06)
  Week 4 | -0.67 (0.09) | -0.72 (0.07) | -0.85 (0.07) | -0.58 (0.07)
  Week 5 | -0.81 (0.10) | -0.79 (0.08) | -1.02 (0.08) | -0.68 (0.08)
  Week 6 | -0.91 (0.11) | -0.99 (0.09) | -1.19 (0.08) | -0.81 (0.09)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare the average effect analysis for brexpiprazole 2 mg/day and 4 mg/day and placebo combined treatment groups at Week 6; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6. The analysis of this key secondary endpoint was conducted if both comparisons of brexpiprazole 4 mg/day vs placebo and brexpiprazole 2 mg/day vs placebo of the primary endpoint were significant. Because only the comparison of brexpiprazole 4 mg/day vs placebo met the threshold in the primary analysis, the following analysis is not part of the formal statistical testing and is descriptive only; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.62 to -0.15]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1269, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.42 to -0.05]
Statistical Analysis 4: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.4449, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.37 to 0.16]

3. Secondary Outcome: Mean Change From Baseline to Week 6 in Personal and Social Performance (PSP) Score.
Description: PSP is a validated clinician-rated scale that measures personal and social functioning in 4 domains: socially useful activities (e.g. work and study), personal and social relationships, self-care, and disturbing and aggressive behaviors. Impairment in each of these domains was rated as absent, mild, manifest, marked, severe, or very severe. These ratings were then converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval, and the rater's judgment to determine the total score within the 10-point interval. Participants with a PSP total score of 71 to 100 were considered to have mild functional difficulty. Scores of 31 to 70 represented manifest disabilities of various degrees and ratings of 1 to 30 indicated minimal functioning that required intense support and/or supervision.
Time Frame: Baseline, Week 3 and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 105 | 170 | 174 | 163
Units on a scale
  Week 3 | 6.97 (0.90) | 6.85 (0.73) | 7.12 (0.71) | 5.80 (0.73)
  Week 6 | 11.73 (1.19) | 10.52 (0.95) | 13.11 (0.94) | 8.52 (0.97)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.59, 95% CI 2-sided [2.02 to 7.17]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1286, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.00, 95% CI 2-sided [-0.58 to 4.59]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0332, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [0.26 to 6.16]

4. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Positive Subscale Score.
Description: PANSS consisted of three subscales: a total of 30 symptom constructs. For each construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS positive subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome). The analysis of secondary endpoints was conducted if both comparisons of brexpiprazole 4 mg/day vs placebo and brexpiprazole 2 mg/day vs placebo of the primary endpoint were significant. Although only the comparison of brexpiprazole 4 mg/day vs placebo met the gatekeeping threshold in the primary analysis, statistical testing for the other doses was reported for information.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -0.93 (0.28) | -1.43 (0.23) | -1.80 (0.23) | -1.25 (0.23)
  Week 2 | -2.54 (0.39) | -2.76 (0.32) | -2.93 (0.32) | -2.56 (0.32)
  Week 3 | -3.94 (0.46) | -3.56 (0.37) | -4.43 (0.37) | -3.34 (0.37)
  Week 4 | -4.83 (0.52) | -4.35 (0.42) | -5.16 (0.41) | -3.93 (0.42)
  Week 5 | -4.80 (0.58) | -4.68 (0.47) | -6.04 (0.46) | -4.33 (0.47)
  Week 6 | -5.63 (0.62) | -5.42 (0.50) | -6.65 (0.50) | -4.95 (0.51)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0166, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-3.08 to -0.31]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.5101, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.86 to 0.93]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.3938, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-2.26 to 0.89]

5. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Negative Subscale Score.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS negative subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -0.31 (0.25) | -0.52 (0.20) | -0.88 (0.20) | -0.40 (0.20)
  Week 2 | -1.27 (0.29) | -1.31 (0.23) | -1.42 (0.23) | -0.79 (0.24)
  Week 3 | -2.06 (0.35) | -1.80 (0.28) | -2.15 (0.28) | -1.18 (0.28)
  Week 4 | -2.56 (0.40) | -2.09 (0.32) | -2.69 (0.32) | -1.67 (0.33)
  Week 5 | -2.71 (0.44) | -2.50 (0.35) | -2.82 (0.35) | -1.74 (0.36)
  Week 6 | -2.92 (0.48) | -2.91 (0.38) | -3.36 (0.38) | -2.14 (0.39)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0231, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.28 to -0.17]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1547, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.83 to 0.29]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.2004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.98 to 0.42]

6. Secondary Outcome: Mean Clinical Global Impression-Improvement (CGI-I) Scale Score at Week 6.
Description: The efficacy of trial medication was rated for each participant using the CGI-I. The study physician would rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at Baseline prior to the first dose of double-blind study medication. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 120 | 180 | 183 | 181
Units on a scale | 3.20 (1.45) | 3.17 (1.34) | 2.95 (1.33) | 3.48 (1.46)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenzel (CMH) row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.78 to -0.20]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0422, Cochran-Mantel-Haenszel; CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.60 to -0.01]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1358, Cochran-Mantel-Haenszel; CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.56 to 0.08]

7. Secondary Outcome: Percentage of Participants With Response at Week 6.
Description: The response rate was defined as reduction of ≥30% from Baseline in PANSS Total Score or CGI-I score of 1 or 2.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
percentage of participants | 43.6 | 38.5 | 49.7 | 31.7
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel; CMH general association test; Relative Risk = 1.54, 95% CI 2-sided [1.20 to 2.00]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1680, Cochran-Mantel-Haenszel; CMH general association test; Relative Risk = 1.22, 95% CI 2-sided [0.92 to 1.62]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0433, Cochran-Mantel-Haenszel; CMH general association test; Relative Risk = 1.35, 95% CI 2-sided [1.02 to 1.79]

8. Secondary Outcome: Percentage of Participants With Discontinuation Rate for Lack of Efficacy at Week 6.
Description: Participants discontinued for lack of efficacy during the trial were reported here.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
percentage of participants | 7.69 | 11.2 | 8.84 | 11.7
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.5202, Cochran-Mantel-Haenszel; CMH general association test; Relative Risk = 0.82, 95% CI 2-sided [0.44 to 1.51]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.9894, Cochran-Mantel-Haenszel; CMH general association test; Relative Risk = 1.00, 95% CI 2-sided [0.55 to 1.85]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.4586, Cochran-Mantel-Haenszel; CMH general association test; Relative Risk = 0.76, 95% CI 2-sided [0.36 to 1.59]

9. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Excited Component (PEC) Score.
Description: The PEC score consisted of five PANSS items: excitement (P4), hostility (P7), tension (G4), uncooperativeness (G8), and poor impulse control (G14). Each of the items were rated on a scale of 1 (absent) to 7 (extreme). The PEC scores ranged from 5 (not present) to 35 (extremely severe).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -0.35 (0.25) | -0.46 (0.21) | -1.01 (0.21) | -0.48 (0.21)
  Week 2 | -0.76 (0.32) | -1.31 (0.26) | -1.21 (0.26) | -0.62 (0.26)
  Week 3 | -1.21 (0.35) | -1.31 (0.28) | -1.81 (0.28) | -0.82 (0.29)
  Week 4 | -1.58 (0.37) | -1.52 (0.29) | -2.12 (0.29) | -1.12 (0.30)
  Week 5 | -1.16 (0.42) | -1.48 (0.34) | -2.27 (0.34) | -0.97 (0.35)
  Week 6 | -1.94 (0.41) | -1.90 (0.33) | -2.86 (0.33) | -1.47 (0.34)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-2.30 to -0.48]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.3559, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.34 to 0.48]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.3646, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.51 to 0.56]

10. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Marder Factor Scores: Positive Symptoms Score.
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The positive factor score is the sum of the 8 components of the positive symptoms scale (range: 8 - best possible outcome to 56 - worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -1.44 (0.29) | -1.77 (0.23) | -1.75 (0.24) | -1.30 (0.24)
  Week 2 | -2.97 (0.39) | -3.10 (0.32) | -3.03 (0.32) | -3.03 (0.32)
  Week 3 | -4.48 (0.47) | -4.09 (0.38) | -4.39 (0.37) | -3.78 (0.38)
  Week 4 | -5.42 (0.53) | -4.93 (0.43) | -5.48 (0.43) | -4.67 (0.44)
  Week 5 | -5.86 (0.58) | -5.35 (0.47) | -6.41 (0.46) | -5.47 (0.47)
  Week 6 | -6.56 (0.66) | -6.26 (0.53) | -7.05 (0.53) | -5.91 (0.54)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1273, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-2.61 to 0.33]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.6400, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.83 to 1.12]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.4423, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-2.32 to 1.01]

11. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Marder Factor Scores: Negative Symptoms Score.
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The negative factor score is the sum of the 7 items of the negative subscale (range: 8 - best possible outcome to 56 - worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -0.70 (0.28) | -0.85 (0.22) | -1.12 (0.23) | -0.66 (0.22)
  Week 2 | -1.71 (0.32) | -1.86 (0.26) | -1.72 (0.26) | -1.38 (0.26)
  Week 3 | -2.55 (0.37) | -2.30 (0.30) | -2.64 (0.30) | -1.83 (0.30)
  Week 4 | -3.21 (0.43) | -2.63 (0.34) | -3.17 (0.34) | -2.16 (0.35)
  Week 5 | -3.35 (0.47) | -3.13 (0.38) | -3.21 (0.37) | -2.24 (0.38)
  Week 6 | -3.55 (0.48) | -3.53 (0.39) | -3.84 (0.39) | -2.55 (0.40)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0194, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.36 to -0.21]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0754, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-2.06 to 0.10]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1080, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-2.22 to 0.22]

12. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Marder Factor Scores: Disorganized Thought Score.
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The disorganized thoughts factor score is the sum of score from the 7 items on the disorganized thoughts subscale (range: 7 - best possible outcome to 49 - worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -0.40 (0.23) | -0.46 (0.19) | -0.78 (0.19) | -0.42 (0.19)
  Week 2 | -1.42 (0.27) | -1.15 (0.22) | -1.37 (0.22) | -0.71 (0.23)
  Week 3 | -2.35 (0.31) | -1.71 (0.25) | -2.32 (0.25) | -1.35 (0.26)
  Week 4 | -2.56 (0.36) | -2.27 (0.29) | -2.83 (0.29) | -1.77 (0.30)
  Week 5 | -2.95 (0.41) | -2.55 (0.33) | -3.42 (0.32) | -2.01 (0.33)
  Week 6 | -3.46 (0.43) | -2.94 (0.35) | -3.98 (0.34) | -2.59 (0.35)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6. Because only the comparison of brexpiprazole 4 mg/day versus placebo met the threshold in the primary analysis, the following analysis is not part for the formal statistical testing and is descriptive only; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-2.34 to -0.43]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.4753, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.31 to 0.61]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.1150, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.96 to 0.21]

13. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Marder Factor Scores: Uncontrolled Hostility and Excitement Score.
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The uncontrolled hostility/excitement factor score is the sum of score from the 4 items on the uncontrolled hostility/excitement subscale (range: 4 - best possible outcome to 28 - worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 4 mg: Brexpiprazole 4 mg tablet once daily for 6 weeks. Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
- Placebo: Placebo tablet once daily for 6 weeks. Participants were titrated to the target dose of placebo over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | 0.03 (0.22) | -0.10 (0.18) | -0.63 (0.18) | -0.21 (0.18)
  Week 2 | -0.15 (0.28) | -0.65 (0.23) | -0.68 (0.23) | -0.13 (0.23)
  Week 3 | -0.46 (0.30) | -0.61 (0.24) | -1.16 (0.24) | -0.19 (0.24)
  Week 4 | -0.74 (0.32) | -0.74 (0.26) | -1.31 (0.25) | -0.39 (0.26)
  Week 5 | -0.34 (0.36) | -0.60 (0.29) | -1.50 (0.29) | -0.22 (0.30)
  Week 6 | -0.90 (0.36) | -0.81 (0.29) | -1.89 (0.29) | -0.64 (0.30)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-2.05 to -0.46]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.6792, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.97 to 0.63]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.5752, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.16 to 0.65]

14. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Marder Factor Scores: Anxiety and Depression Score.
Description: Retrospective factor analyses have been performed in recent decades using scores for the 30 individual PANSS items to categorize symptoms into 5 dimensions. Collectively, these dimensions are referred to as the PANSS Marder Factor scores and include positive symptoms score, negative symptoms score, thought score, uncontrolled hostility/excitement, anxiety depression score. The anxiety/depression factor score is the sum of score from the 4 items on the anxiety/depression subscale (range: 4 - best possible outcome to 28 - worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Number analyzed (Participants) | 117 | 179 | 181 | 180
Units on a scale
  Week 1 | -1.18 (0.22) | -1.10 (0.18) | -1.26 (0.18) | -0.96 (0.18)
  Week 2 | -1.86 (0.27) | -1.91 (0.22) | -1.60 (0.22) | -1.47 (0.22)
  Week 3 | -2.43 (0.28) | -2.10 (0.23) | -2.24 (0.23) | -1.97 (0.23)
  Week 4 | -2.85 (0.29) | -2.70 (0.23) | -2.93 (0.23) | -2.60 (0.23)
  Week 5 | -2.93 (0.31) | -2.87 (0.25) | -3.09 (0.25) | -2.69 (0.26)
  Week 6 | -3.57 (0.30) | -3.62 (0.24) | -3.78 (0.24) | -2.93 (0.24)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Placebo; Statistical analysis to compare brexpiprazole 4mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0104, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.51 to -0.20]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0373, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.35 to -0.04]
Statistical Analysis 3: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1mg/day and placebo was performed at Week 6; Test type: Superiority or Other; p = 0.0890, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.39 to 0.10]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 30 (+2) days after the last dose of study medication.
Description: A serious adverse event (SAE) was an untoward medical occurrence that resulted in death or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or a new problem experienced by a participant when enrolled in a trial whether or not it was considered drug related by study physician.
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/120 | 4/186 | 4/184 | 10/184
Other Adverse Events (participants affected / at risk) | 37/120 | 65/186 | 66/184 | 71/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1 mg (N=120) | Brexpiprazole 2 mg (N=186) | Brexpiprazole 4 mg (N=184) | Placebo (N=184)
Irritability (General disorders) | 0 | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 2 | 1 | 1
Schizophrenia (Psychiatric disorders) | 1 | 2 | 3 | 8
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1 mg (N=120) | Brexpiprazole 2 mg (N=186) | Brexpiprazole 4 mg (N=184) | Placebo (N=184)
Dyspepsia (Gastrointestinal disorders) | 7 | 7 | 6 | 6
Akathisia (Nervous system disorders) | 5 | 9 | 12 | 13
Headache (Nervous system disorders) | 9 | 20 | 19 | 27
Agitation (Psychiatric disorders) | 10 | 16 | 13 | 13
Insomnia (Psychiatric disorders) | 15 | 25 | 28 | 27
Schizophrenia (Psychiatric disorders) | 4 | 6 | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No